CLINICAL TRIAL: NCT06577207
Title: Pattern and Outcome of Children Admitted in Emergency Unit of Assuit Children University Hospital
Brief Title: Pattern and Outcome of Children Admitted in Emergency Unit of Assuit Children University Hospital Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ereeny louiz Azmy Sorieal, physician, Assiut University
Other Study IDs: children in Emergency Unit
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Emergency Medicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Initial investigations for all cases — Initial investigations for all cases: 1. Pulse oximetry. 2. Complete blood count. 3. Electrolytes. 4. Kidney function test. 5. Random blood glucose 6. Other investigations ordered for certain cases according to clinical manifestation & previous findings > Lines of treatment will be recorded

SUMMARY:
In the present work, we aim to

1. Describe the pattern of patients admitted to Emergency unite at Assiut University Child Hospital (AUCH) and classify them according to age ,distribution ,most common presenting complain, effect of seasonal variation on causes of admission ,prognosis till discharge of the patient to home or refer him to specific unit in pediatric hospital and associated chronic disease.
2. Describe factors affecting mortality rate

DETAILED DESCRIPTION:
Emergency department (ED) is the essential and important front line of medical care provided by the hospital. Child mortality rates remain high globally; mortality rate is a reflection of the severity of illness and the quality of treatment of patients in pediatric emergency departments . In Africa, the childhood mortality rate is 92 per 1000 live births which are 15 times more than that of well-resourced countries. In pediatric departments, early child mortality is commonly caused by preventable and reversible diseases, so urgent treatment and resuscitation are required to avoid poor outcomes . Overcrowding in ED has also been a global urgent problems , overcrowded could be brought by multiple factors as a facility with rapid diagnostic modalities and early initiation of therapy and patients can expect a higher possibility to be admitted to the hospital by the ED attendant . Early identification and treatment of pneumonia, sepsis, heart failure (secondary to anemia), acute respiratory tract infections, and diarrheal diseases has been shown to reduce childhood mortality in acute pediatric hospitals. Critical clinical issues, such as shortness of breath, fast breathing and fever with seizure are some of the preventable causes contributing to childhood mortality. Effective intervention and good emergency care and classification of children requires effort and coordination starting from the bedside up to the governmental level .

ELIGIBILITY:
Inclusion Criteria:

* All patients from 28 day till 18 years who will be admitted to emergency unite at (AUCH) during duration of the study,data of the patients will be collected in the form of :

  * Full history taking:

    1. Personal history: (age, sex, gestational age), residence and socioeconomic status.
    2. Cause of admission and clinical characteristic of patients (medical or surgical condition).
    3. Triage and acuity : rapidly screening of sick children in order to identify: • those with emergency signs, who require immediate emergency treatment; • those with priority signs, who are at higher risk of dying.

       These children should be assessed without unnecessary delay. • non-urgent cases, who have neither emergency nor priority signs. Emergency signs include: obstructed or absent breathing, severe respiratory distress, central cyanosis, signs of shock, coma, convulsions, signs of severe dehydration . The priority signs include: any sick child aged < 2 months, very high temperature, severe pallor, history of poisoning, severe pain, restless or continuously irritable, edema of both feet
    4. Associated symptoms of different systems involved.
    5. Provisional diagnosis.
    6. 1 st admission or not
    7. Referring center , time and seasonal variation to detect most peak area and months
    8. Fate
  * Complete physical examination: Including body temperature , respiratory rate, heart rate, pallor, weight loss, and evidence of dehydration. Chest, cardiac , abdominal and neurological examination.
  * Investigations and Imaging: Initial investigations for all cases: 1. Pulse oximetry. 2. Complete blood count. 3. Electrolytes. 4. Kidney function test. 5. Random blood glucose 6. Other investigations ordered for certain cases according to clinical manifestation & previous findings > Lines of treatment will be recorded
  * Patients will be followed during their stay in ER and till discharge patient to home or refer him to specific unit in pediatric hospital with monitoring of factors affecting their prognosis.

Exclusion Criteria:

1. Neonates
2. patients which their age are more than 18 years
3. Patients which have recent trauma

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The present study is a cross-sectional study.study will be carried out on patients admitted to Emergency unite at Assiut University Child Hospital (AUCH) .An informed consent will be obtained from all patients. The study will be conducted in Assiut university child hospital, during the period from Jan 2025 to Jan 2026 .The purpose and nature of the study will be explained to all patients.
  At least 94 patients will be included in the present study. The sample size was calculated using Epi-info version 7software,Based on previous studies, the confidence limits of 5% , a confidence level =80% ,and the rate of pediatric patients emergency admission as 50% , and allocation ratio of 1.
Sampling Method: Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
classification of pediatric patient in emergency room | baseline
  classification of pediatric patient in emergency room according to age distribution
  ,most common presenting complain, effect of seasonal variation on causes of admission ,prognosis till discharge of the patient to home or refer him to specific unit in pediatric hospital and associated chronic disease.

SECONDARY OUTCOMES:
search for factors affect mortality rate | baseline
  search for factors affect mortality rate

REFERENCES:
- [Background] Rothman RE, Irvin CB, Moran GJ, Sauer L, Bradshaw YS, Fry RB Jr, Josephson EB, Ledyard HK, Hirshon JM; Public Health Committee of the American College of Emergency Physicians. Respiratory hygiene in the emergency department. Ann Emerg Med. 2006 Nov;48(5):570-82. doi: 10.1016/j.annemergmed.2006.05.018. Epub 2006 Aug 23. PMID 17052558
- [Background] Liu L, Oza S, Hogan D, Perin J, Rudan I, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of child mortality in 2000-13, with projections to inform post-2015 priorities: an updated systematic analysis. Lancet. 2015 Jan 31;385(9966):430-40. doi: 10.1016/S0140-6736(14)61698-6. Epub 2014 Sep 30. PMID 25280870